CLINICAL TRIAL: NCT07086040
Title: Effects of Rhythmic Auditory Stimulation Therapy on Upper-Limb Movements, Function, and Quality of Life in Patients With Schizophrenia: Randomized Controlled Trials
Brief Title: Effects of RAS in SZ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shu-Mei Wang (Other)
Responsible Party: Sponsor-Investigator, Shu-Mei Wang, Dr., National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAS in SZ
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia and Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SZ patients receiving second-generation antipsychotics + RAS (Experimental): SZ patients receiving second-generation antipsychotics: Provision of upper-limb movement training with the aid of RAS
  Interventions: Behavioral: RAS incorporated in upper-limb movement training
- SZ patients receiving second-generation antipsychotics + no RAS (Active Comparator): SZ patients receiving second-generation antipsychotics: Provision of upper-limb movement training without the aid of RAS
  Interventions: Behavioral: Upper-limb movement training
- SZ patients receiving first-generation antipsychotics + RAS (Experimental): SZ patients receiving first-generation antipsychotics: Provision of upper-limb movement training with the aid of RAS
  Interventions: Behavioral: RAS incorporated in upper-limb movement training
- SZ patients receiving first-generation antipsychotics + no RAS (Active Comparator): SZ patients receiving first-generation antipsychotics: Provision of upper-limb movement training without the aid of RAS
  Interventions: Behavioral: Upper-limb movement training

INTERVENTIONS:
Behavioral: RAS incorporated in upper-limb movement training — RAS will be metronome beat sound with different tempi and will be incorporated in upper-limb movement training, which will last for 40 minutes per session for a total of 21 sessions.
  Arms: SZ patients receiving first-generation antipsychotics + RAS; SZ patients receiving second-generation antipsychotics + RAS
Behavioral: Upper-limb movement training — Upper-limb movement training will last for 40 minutes per session for a total of 21 sessions.
  Arms: SZ patients receiving first-generation antipsychotics + no RAS; SZ patients receiving second-generation antipsychotics + no RAS

SUMMARY:
The two main groups of medicated patients with schizophrenia (SZ) are those receiving second-generation antipsychotics and those receiving first-generation antipsychotics. The purpose of this research project is to target each patient group to examine effects of rhythmic auditory stimulation (RAS) on upper-limb movements in medicated SZ patients in a 6-month follow-up period.

The main questions of this project are:

1. Does RAS reduce severity of upper-limb bradykinesia (slow movements) and dyskinesia (repetitive and involuntary movements) after intervention, at 3-month follow-up and 6-month follow-up in SZ patients receiving second-generation antipsychotics? and
2. Does RAS reduce severity of upper-limb bradykinesia and dyskinesia after intervention, at 3-month follow-up and 6-month follow-up in SZ patients receiving first-generation antipsychotics?

Researchers will compare upper-limb movement training with the aid of RAS to upper-limb movement training without the aid of RAS to see if RAS works to improve upper-limb movements in SZ patients. Participants will:

1. Undergo an interview and movement tests and fill out questionnaires before and after the movement training program and at 3-month follow-up and 6-month follow-up; and
2. Receive movement training for 40 minutes per session for a total of 21 sessions.

ELIGIBILITY:
[For SZ patients]

Inclusion Criteria:

* A diagnosis of schizophrenia or schizoaffective disorder
* Between 18 to 60 years old
* Keeping the same antipsychotics and the same dosage at least 4 weeks right before joining the study
* A Edinburgh Handedness Inventory score of > 60
* A Montreal Cognitive Assessment score of ≥ 24

Exclusion Criteria:

* Substance abuse or drug abuse
* Neurological diseases or medical conditions that affect upper-limb movements and hearing
* Other psychiatric diagnoses in addition to a diagnosis of schizophrenia or schizoaffective disorder

[For healthy participants]

Inclusion Criteria:

* Between 18 to 60 years old
* A Edinburgh Handedness Inventory score of > 60
* A Montreal Cognitive Assessment score of ≥ 24

Exclusion Criteria:

* Substance abuse or drug abuse
* Neurological diseases or medical conditions that affect upper-limb movements and hearing
* Psychiatric diagnoses
* Taking psychotropic medications
* Presence of first-degree relatives or siblings with diagnoses of psychiatric diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Purdue pegboard test | Up to 1 week right before the 1st session of the intervention
  A larger value (the number of inserted pins) means a faster movement.
Purdue pegboard test | Up to 1 week right after the last session of the intervention
  A larger value (the number of inserted pins) means a faster
Purdue pegboard test | After three months following the last session of the intervention
  A larger value (the number of inserted pins) means a faster movement.
Purdue pegboard test | After six months following the last session of the intervention
  A larger value (the number of inserted pins) means a faster movement.
Box and Block Test | Up to 1 week right before the 1st session of the intervention
  A larger value (the number of blocks) means a faster movement.
Box and Block Test | Up to 1 week right after the last session of the intervention
  A larger value (the number of blocks) means a faster movement.
Box and Block Test | After three months following the last session of the intervention
  A larger value (the number of blocks) means a faster movement.
Box and Block Test | After six months following the last session of the intervention
  A larger value (the number of blocks) means a faster movement.
Extrapyramidal Symptom Rating Scale | Up to 1 week right before the 1st session of the intervention
  A larger score means more severe bradykinesia
Extrapyramidal Symptom Rating Scale | Up to 1 week right after the last session of the intervention
  A larger score means more severe bradykinesia
Extrapyramidal Symptom Rating Scale | After three months following the last session of the intervention
  A larger score means more severe bradykinesia
Extrapyramidal Symptom Rating Scale | After six months following the last session of the intervention
  A larger score means more severe bradykinesia
Abnormal Involuntary Movement Scale | Up to 1 week right before the 1st session of the intervention
  A larger score means more severe dyskinesia
Abnormal Involuntary Movement Scale | Up to 1 week right after the last session of the intervention
  A larger score means more severe dyskinesia
Abnormal Involuntary Movement Scale | After three months following the last session of the intervention
  A larger score means more severe dyskinesia
Abnormal Involuntary Movement Scale | After six months following the last session of the intervention
  A larger score means more severe dyskinesia

SECONDARY OUTCOMES:
Jebsen-Taylor Hand Function Test | Up to 1 week right before the 1st session of the intervention
  A larger value (the time for completing the task) of each task means a slower movement.
Jebsen-Taylor Hand Function Test | Up to 1 week right after the last session of the intervention
  A larger value (the time for completing the task) of each task means a slower movement.
Jebsen-Taylor Hand Function Test | After three months following the last session of the intervention
  A larger value (the time for completing the task) of each task means a slower movement.
Jebsen-Taylor Hand Function Test | After six months following the last session of the intervention
  A larger value (the time for completing the task) of each task means a slower movement.
Averaged weekly working hours | Up to 1 week right before the 1st session of the intervention
  A larger value (working hours) means higher working function.
Averaged weekly working hours | Up to 1 week right after the last session of the intervention
  A larger value (working hours) means higher working function.
Averaged weekly working hours | After three months following the last session of the intervention
  A larger value (working hours) means higher working function.
Averaged weekly working hours | After six months following the last session of the intervention
  A larger value (working hours) means higher working function.
The short version of the World Health Organization Quality of Life questionnaire | Up to 1 week right before the 1st session of the intervention
  A larger score means higher quality of life.
The short version of the World Health Organization Quality of Life questionnaire | Up to 1 week right after the last session of the intervention
  A larger score means higher quality of life.
The short version of the World Health Organization Quality of Life questionnaire | After three months following the last session of the intervention
  A larger score means higher quality of life.
The short version of the World Health Organization Quality of Life questionnaire | After six months following the last session of the intervention
  A larger score means higher quality of life.
Positive and Negative Syndrome Scale | Up to 1 week right before the 1st session of the intervention
  A larger score means more severe psychotic symptoms.
Positive and Negative Syndrome Scale | Up to 1 week right after the last session of the intervention
  A larger score means more severe psychotic symptoms.
Positive and Negative Syndrome Scale | After three months following the last session of the intervention
  A larger score means more severe psychotic symptoms.
Positive and Negative Syndrome Scale | After six months following the last session of the intervention
  A larger score means more severe psychotic symptoms.
The Montreal Cognitive Assessment | Up to 1 week right before the 1st session of the intervention
  A larger score means higher cognition.
The Montreal Cognitive Assessment | Up to 1 week right after the last session of the intervention
  A larger score means higher cognition.
The Montreal Cognitive Assessment | After three months following the last session of the intervention
  A larger score means higher cognition.
The Montreal Cognitive Assessment | After six months following the last session of the intervention
  A larger score means higher cognition.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No